CLINICAL TRIAL: NCT07366918
Title: Comparison of the Efficacy of Perineal and Intravaginal Electrical Stimulation in Women With Idiopathic Overactive Bladder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Necmettin Yildiz, Professor Doctor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: E-60116787-020-728459
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Urinary Bladder, Overactive
Keywords: Idiopathic overactive bladder; Urinary incontinence; perineal electrical stimulation; Intravaginal electrical stimulation
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BT + Intravaginal ES (Experimental): In this group, IVES will be administered in addition to BT. IVES will be performed in the lithotomy position using a vaginal probe and a stimulation device (Enraf Nonius Myomed 632). IVES will be performed three days a week for 20 minutes per day for 8 weeks, totaling 24 sessions. Stimulation parameters will be a frequency of 10 Hz, a 5-10 second work-rest cycle, and a 100 ms pulse width. A symmetrical biphasic pulse wave can be delivered in the range of 1-100 mA (based on the patient's discomfort level feedback) . IVES sessions will be performed by a physical medicine and rehabilitation physician.
  Interventions: Other: Bladder Training + Intravaginal ES
- BT + Perineal ES (Experimental): Perineal ES will be administered in the lithotomy position using a combined electrotherapy stimulation device with surface electrodes (Enraf Nonius Myomed 632). Perineal ES will be administered 20 minutes per day, 3 days per week, for 8 weeks, for a total of 24 sessions. Stimulation parameters will be 10 Hz frequency, 5-10 s work-rest cycle, and 100 µs pulse width. A symmetrical biphasic current wave can be delivered in the 1-100 mA range (depending on the patient's discomfort level feedback). In this application, five 2 cm diameter surface electrodes will be used: four electrodes symmetrically in the perianal region and one electrode (ground-neutral electrode) on the leg. Patients will not perform voluntary contractions during ES. Surface electrodes will be used individually for each patient. Perineal ES sessions will be performed by a physical medicine and rehabilitation physician
  Interventions: Other: Bladder Training + Perineal ES
- Bladder Training (BT) (Active Comparator): All women will be informed about BT, which consists of four stages lasting 30 minutes. A written brochure will then be provided as a program that can be implemented at home. In the first stage, women will be informed about the location of the BT, pelvic anatomy, and pathophysiology. Following this informational session, they will be demonstrated how to squeeze the BT at least once using digital palpation techniques to suppress urgency. In the second stage, which includes urgency suppression strategies, the aim is to delay urination, inhibit detrusor contraction, and prevent urgency by squeezing the BT several times in a row, taking deep breaths, focusing on another task for a while, and self-motivating themselves. In the third stage, a timed voiding program will be initiated. This will be carried out in two steps: timed voiding and increasing the time between voids by keeping a voiding diary. In the final stage, women will be encouraged to continue BT
  Interventions: Other: BT

INTERVENTIONS:
Other: Bladder Training + Intravaginal ES — IVES will be performed in the lithotomy position using a vaginal probe and a stimulation device . IVES will be performed three days a week for 20 minutes per day for 8 weeks, totaling 24 sessions. Stimulation parameters will be a frequency of 10 Hz, a 5-10 second work-rest cycle, and a 100 ms pulse width. A symmetrical biphasic pulse wave can be delivered in the range of 1-100 mA (based on the patient's discomfort level feedback).
  Arms: BT + Intravaginal ES
Other: BT — A written brochure will then be provided as a program that can be implemented at home. In the first stage, women will be informed about the location of the BT, pelvic anatomy, and pathophysiology. Following this informational session, they will be demonstrated how to squeeze the BT at least once using digital palpation techniques to suppress urgency. In the second stage, which includes urgency suppression strategies, the aim is to delay urination, inhibit detrusor contraction, and prevent urgency by squeezing the BT several times in a row, taking deep breaths, focusing on another task for a while, and self-motivating themselves. In the third stage, a timed voiding program will be initiated. This will be carried out in two steps: timed voiding and increasing the time between voids by keeping a voiding diary. In the final stage, women will be encouraged to continue BT
  Arms: Bladder Training (BT)
Other: Bladder Training + Perineal ES — Perineal ES will be administered in the lithotomy position using a combined electrotherapy stimulation device with surface electrodes. Perineal ES will be administered 20 minutes per day, 3 days per week, for 8 weeks, for a total of 24 sessions. Stimulation parameters will be 10 Hz frequency, 5-10 s work-rest cycle, and 100 µs pulse width. A symmetrical biphasic current wave can be delivered in the 1-100 mA range (depending on the patient's discomfort level feedback). In this application, five 2 cm diameter surface electrodes will be used: four electrodes symmetrically in the perianal region and one electrode (ground-neutral electrode) on the leg. Patients will not perform voluntary contractions during ES. Surface electrodes will be used individually for each patient. Perineal ES sessions will be performed by a physical medicine and rehabilitation physician.
  Arms: BT + Perineal ES

SUMMARY:
The investigators conducted a prospective, randomized double-blind, placebo-controlled study based on a placebo technique to evaluate the efficacy of IVES vs perineal ES in women with idiopathic OAB.

The main questions aimed to be answered are:

Is Intravaginal Electrical Stimulation (IVES) or perineal ES more effective on clinical parameters related to incontinence and quality of life in women with idiopathic overactive bladder (OAB)? Participants (n:63) with idiopathic OAB who meet the exclusion and inclusion criteria will be divided into 3 groups using a randomization table. The first group will receive IVES and bladder training (n:21), second group will receive perineal ES and bladder training (n:21) and third group will receive bladder training (n=21) . Measurements will be performed twice in total, before and at the end of treatment (8th week).

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18 with a clinical diagnosis of idiopathic OAB
* Intolerant or unresponsive to antimuscarinic or oral β3 adrenoceptor agonist (mirabegron) medications and not using them for at least 4 weeks
* Ability to understand the procedures, advantages, and potential side effects
* Ability to provide written, informed consent
* Pelvic floor muscle (PFM) strength of 3/5 or higher (modified Oxford scale, minimum: 0 - maximum: 5)

Exclusion Criteria:

* Women with pure stress urinary incontinence
* History of conservative treatment for OAB within the last 6 months (MI, IVES, perineal ES, etc.)
* Pregnant or planning to become pregnant at the time of the study
* Diagnosis of vaginal infection, urinary tract infection, or cancer
* Women with urinary incontinence within the last 3 months Those who have undergone urogynecological surgery
* Those with genital area disorders that may preclude the use of a vaginal probe or perineal electrode
* Those diagnosed with stage 2 or higher according to the Pelvic Organ Prolapse Assessment (POP-Q)
* Those with a pacemaker or implanted defibrillator
* Those with neurogenic bladder or a history of neurological disease
* Those with a urine residual of more than 100 ml detected by ultrasound (using an ultrasound device)
* Those with allergies to condoms or lubricating gels used with a vaginal probe or perineometer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 63 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in incontinence episodes | Change from baseline Improvement in incontinence episodes at the 8th week after the treatment
  Reduction in incontinence episodes will be collected. Women with ≥50% reduction in incontinence episodes will be considered positive responders

SECONDARY OUTCOMES:
The severity of incontinence | Change from baseline the severity of incontinence at the 8th week after the treatment
  The 24-hour pad test was carried out to evaluate the severity of incontinence
Symptom severity | Change from baseline symptom severity at the 8th week after the treatment
  Overactive Bladder Questionnaire (OAB-V8) will be used to evaluate symptom severity in women with OAB in the study. The OAB-V8 consists of 8 questions in which patients can be classified as symptom severity: none (0), very little (1), a little (2), quite a few (3), very (4), and too many (5). The total score ranges from 0-40.
Frequency of voiding, nocturia, number of pads | Change from baseline Frequency of voiding, nocturia, number of pads at the 8th week after the treatment
  The frequency of voiding, nocturia, and the number of pads used will be collected from the 3-day bladder diary.
The Quality of Life | Change from baseline the Quality of Life at the 8th week after the treatment
  The Quality of Life-Incontinence Impact Questionnaire (IIQ7) will be used to assess specific QoL related to incontinence
Anxiety and Depression level | Change from baseline anxiety and Depression level at the 8th week after the treatment
  The Hospital Anxiety and Depression Scale (HAD), validated and reliability tested in Turkey in 1987, assesses levels of anxiety and depression. It comprises 14 questions, seven for anxiety and seven for depression, scored on a four-point Likert scale. Scores are summed for each subscale: questions 1, 3, 5, 7, 9, 11, and 13 for anxiety, and questions 2, 4, 6, 8, 10, 12, and 14 for depression. In Turkey, cutoff scores are 10/11 for anxiety and 7/8 for depression, indicating risk.
Assessment of sexual functions Assessment of sexual functions | Change from baseline assessment of sexual functions at the 8th week after the treatment
  In the evaluation of sexual function, the Female Sexual Function Index questionnaire is used, consisting of 19 questions assessing six main factors: sexual desire, arousal, lubrication, orgasm, satisfaction, and pain/discomfort. The highest possible total raw score is 95, while the lowest is 4. After multiplying the coefficients, the highest score is 36, and the lowest is 2. Impact coefficients used for scoring are: 0.6 for sexual desire, 0.3 for arousal and lubrication, and 0.4 for orgasm, satisfaction, and pain/discomfort. An Female Sexual Function Index score below 26.55 is indicative of sexual dysfunction
Cure and improvement rates | Change from baseline cure and improvement rates at the 8th week after the treatment
  Cure and improvement rates will be recorded in all groups at the end-of-treatment assessments. Values under 1.3 g in the 24-hour pad test will be considered as "cure", while a 50% or greater reduction in wet weight compared to baseline measurements at the end of treatment will be considered as "improvement
Treatment Satisfaction Level | Change from baseline Treatment Satisfaction Level at the 8th week after the treatment
  At the end of the treatment, participants will be asked to evaluate their satisfaction level with the administered treatment using a Likert scale ranging from 1 to 5 (5=very satisfied, 4=satisfied, 3=neither satisfied nor dissatisfied, 2=dissatisfied, 1=very dissatisfied).
Pelvic Floor Muscle (PFM) Strength | Change from baseline Pelvic Floor Muscle (PFM) Strength at the 8th week after the treatment
  PFM strength will be assessed using the Peritron 9300 device
Side Effects | 8th week
  All patients will be questioned about side effects such as numbness, fatigue, pain in and around the pelvic floor muscle, and changes and discomfort associated with defecation, drowsiness, headache, fatigue, and asthenia.

CONTACTS AND LOCATIONS:
Overall Officials: Necmettin YILDIZ Prof., Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)